CLINICAL TRIAL: NCT00670059
Title: Pre-Implantation Genetic Screening in Women Under the Age of 36 With Single-Embryo Transfer
Brief Title: Pre-Implantation Genetic Screening in Women Under the Age of 36 Years With Single Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the first prespecified interim analysis
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Staessen Catherine Ph.D., UZBrussel
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SET study
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Live Birth Delivery Rate
Keywords: Single embryo transfer/ aneuploidy screening
MeSH Terms: interventions — Single Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): group: single embryo transfer without aneuploidy screening
  Interventions: Genetic: single embryo transfer without aneuploidy screening
- B (Experimental): group: single embryo transfer with aneuploidy screening
  Interventions: Genetic: single embryo transfer with aneuploidy screening

INTERVENTIONS:
Genetic: single embryo transfer without aneuploidy screening — without aneuploidy testing for the chromosomes XY, 13, 16, 18, 21, 22
  Arms: A
Genetic: single embryo transfer with aneuploidy screening — with aneuploidy testing for the chromosomes XY, 13, 16, 18, 21, 22
  Arms: B

SUMMARY:
BACKGROUND: Single-embryo transfer is a well-accepted strategy to avoid multiple pregnancies in an assisted reproductive technology programme. The selection of the embryo with the highest implantation potential is a crucial step. Besides the morphological quality and embryo kinetics up to the blastocyst stage, pre-implantation genetic screening (PGS) of aneuploidy has been advocated as an adjuvant approach by which to select the right embryo for transfer.

METHODS: Couples with a female partner younger than 36 years were randomly assigned to undergo transfer of a single blastocyst in a cycle with or without PGS using fluorescence in situ hybridization for the chromosomes X, Y, 13, 16, 18, 21 and 22.

DETAILED DESCRIPTION:
Study design Between October 2004 and December 2006, ovulatory women undergoing infertility treatment were asked to participate in this RCT subject to the following inclusion criteria: maternal age below 36 years, need for ICSI and having motile sperm (sperm parameters: more than 1 x 106 sperm cells/ml) and both partners having a normal karyotype. Following written informed consent, eligible couples were randomly assigned to ICSI followed by blastocyst transfer either with or without PGS on the eight-cell stage embryo. Randomization was performed at the outpatient clinic, and each patient could be included only once. The consent form mentioned that patients allocated to PGS group would agree to donate embryos for research if these were chromosomally abnormal or unsuitable for transfer or cryopreservation. The study was approved by the Ethics Committee of the University Hospital. The patients were aware of the treatment allocation and were informed at the moment of transfer concerning the chromosomal abnormalities observed and about the morphological quality of the embryos.

Ovarian stimulation, oocyte retrieval and embryo culture Controlled ovarian hyperstimulation was carried out in an antagonist protocol using recombinant FSH combined with a GnRH antagonist (ganirelix, Orgalutran, NV Organon) (Kolibianakis et al., 2004) or an agonist protocol, using GnRH analogues for pituitary desensitisation (buserilin, Suprefact; Hoechst, Frankfurt, Germany), combined with human menopausal gonadotrophins (hMG)(Menopur, Ferring Pharmaceuticals A/S, Copenhagen, Denmark) or recombinant FSH (Puregon, NV Organon, Oss, The Netherlands)(Van de Velde et al., 1998). Final oocyte maturation was induced by the administration of 10,000 IU of HCG. Transvaginal ultrasound-guided oocyte retrieval was scheduled 36 h after HCG administration. ICSI was used to fertilize the oocytes. Sperm preparation, in vitro fertilization, intracytoplasmic sperm injection procedures and embryo culture were carried out as described by Van Landuyt et al. (2005).

Assessment of fertilization and embryo evaluation Fertilization was assessed as the number of 2PN zygotes per COC retrieved. Embryo evaluation was performed on days 2 and 3 by recording number of blastomeres and percentage of fragmentation. Grade A embryos were defined as embryos without anucleate fragments. Grade B embryos had blastomeres of equal or unequal sizes, with a maximum of 20 % of the volume of the embryo filled with anucleate fragments. In grade C embryos, anucleate fragments were present in 20-50 % of the volume of the embryo. Grade D embryos had more than 50% of the volume of the embryo filled with anucleate fragments. The embryos were evaluated daily until day 5. On day 5, the embryos were classified into arrested embryos showing no signs of compaction on day 5, compacting embryos (C1-C2), early blastocysts (Bl1-Bl2) and expanding blastocysts (Bl3-Bl7) according to the classification proposed by Gardner and Schoolcraft (1999). Embryos were considered for transfer at day 5 only from the compacting stage on. In both groups, supernumerary embryos were cryopreserved on day 5 or 6.

Embryo biopsy Embryos of grade A, B or C with at least five blastomeres were biopsied (Joris et al., 2003) in the morning of day 3 after ICSI. These selection criteria to decide whether an embryo was suitable for biopsy were the same as those used to decide whether an embryo was transferable on day 3 in the regular ICSI programme without PGD. Before biopsy of one blastomere, the blastomeres were checked for the presence of nuclei. If consequently no nuclear material was found during fixation, a second blastomere was removed. Embryo biopsy was carried out in HEPES-buffered medium under oil using laser technology (Fertilase) as was earlier described in detail (Staessen et al., 2004).

Spreading of the interphase nuclei and FISH procedure Using a mouth pipette, the individual blastomeres were first rinsed in medium and then transferred to a 1 µl droplet of 0.01 N HCl/ 0.1% Tween 20 solution (Coonen et al., 1994) on a Superfrost Plus glass slide (Kindler GmbH, Freiburg, Germany). A two-round FISH procedure was performed allowing us to detect the chromosomes X, Y, 13, 18, 21 (round 1) and 16, 22 (round 2) as was previously described in detail (Staessen et al., 2004).

FISH scoring criteria The specific FISH signals detected in a given blastomere were interpreted as follows: (i) a blastomere was considered to be diploid when the two gonosomes and two chromosome 13-, 16-, 18-, 21- and 22 specific signals were present; (ii) a blastomere was considered to be haploid, triploid or tetraploid when respectively one, three or four signals for the investigated chromosomes were present; (iii) a blastomere was considered to be aneuploid when an extra (trisomic) or missing (monosomic) signal for one chromosome was observed, in the presence of two signals for the remaining chromosomes analysed; (iv) a blastomere was considered as combined abnormal when it was neither diploid nor haploid, triploid, tetraploid or aneuploid. After FISH analysis, only embryos found to be chromosomally normal in the corresponding biopsied blastomere were transferred on day 5. FISH analysis was performed by experienced cytogeneticists trained in cytogenetics and FISH analysis. The results of the first and second round were analysed by two observers using a Zeiss Axioplan 2 fluorescence microscope.

Embryo transfer In the PGS group the transfer was performed on day 5 if at least one compacting embryo or early blastocyst was obtained from the embryos found to be genetically normal. In the control group the transfer was also performed if at least one compacting embryo or early blastocyst was obtained on day 5; 4 embryo transfers were performed on day 3.

Pregnancy A biochemical pregnancy was defined as two consecutive positive rising (> 15IU/ml) serum hCG levels. A preclinical miscarriage was defined as two consecutive positive rising (> 15IU/ml) serum hCG levels, but no FHB at least 6 weeks post embryo transfer. A clinical pregnancy was defined as an intrauterine gestational sac with positive foetal heart activity seen at ultrasonography performed at least 6 weeks post-embryo transfer. A miscarriage was defined as a pregnancy loss before 20 weeks of gestation. The live birth delivery rate was defined as the number of live birth deliveries expressed per 100 initiated cycles, aspiration cycles or embryo transfer cycles (Zeghers-Hochschild et al., 2006).

Endpoint The primary outcome was live birth delivery rate. Statistical analysis Analysis was performed according to the intention to treat. For descriptive statistics, we used means±SD. Continuous variables were analyzed by the t-test for independent samples. Categorical variables were analyzed by chi-square test. All tests were two-sided, and a P value of less than 0.05 was considered to indicate statistical significance. Using group sequential methods, we calculated that the enrolment of 447 patients in each group would give the study a statistical power of 80% to detect an absolute difference of 10% in the delivery rate between the groups at an alpha level of 0.05 with the use of a two-sided z-test.

ELIGIBILITY:
Inclusion Criteria:

* ovulatory women undergoing infertility treatment
* maternal age below 36 years
* need for ICSI
* motile sperm: more than 1x1000000 sperm cells/ml
* both having a normal karyotype

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
live born delivery rate | at birth of the child

SECONDARY OUTCOMES:
Number of pregnancies obtained with or without pre-implantation genetic screening | positive HCG

CONTACTS AND LOCATIONS:
Locations (1):
- Staessen C, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Staessen C, Platteau P, Van Assche E, Michiels A, Tournaye H, Camus M, Devroey P, Liebaers I, Van Steirteghem A. Comparison of blastocyst transfer with or without preimplantation genetic diagnosis for aneuploidy screening in couples with advanced maternal age: a prospective randomized controlled trial. Hum Reprod. 2004 Dec;19(12):2849-58. doi: 10.1093/humrep/deh536. Epub 2004 Oct 7. PMID 15471934
- [Derived] Staessen C, Verpoest W, Donoso P, Haentjens P, Van der Elst J, Liebaers I, Devroey P. Preimplantation genetic screening does not improve delivery rate in women under the age of 36 following single-embryo transfer. Hum Reprod. 2008 Dec;23(12):2818-25. doi: 10.1093/humrep/den367. Epub 2008 Oct 17. PMID 18930977